CLINICAL TRIAL: NCT01064024
Title: A Double Blind, Randomized, Parallel Controlled Study to Evaluate the Safety and Efficacy of Phenazopyridine Hydrochloride Tablets, USP 200 mg vs. Placebo as a Urinary Analgesic for Short Term Treatment in Female Subjects Suffering From Pain or Burning When Passing Urine Associated With Uncomplicated Urinary Tract Infections (uUTI)
Brief Title: Evaluate the Safety and Efficacy of Phenazopyridine Hydrochloride Tablets, USP 200 mg vs. Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Oxford Pharmaceutical Resources, Inc. (Industry); Sristek Clinical Research Solutions Limited (Industry); Biostudy Solutions, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-PHN-001
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pain; Urinary Tract Infections
Keywords: uUTI; Pain or burning associated with Uncomplicated Urinary Tract Infections
MeSH Terms: conditions — Pain; Urinary Tract Infections | interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenazopyridine Hydrochloride Tablets, USP 200 mg (Active Comparator)
  Interventions: Drug: Phenazopyridine Hydrochloride
- Placebo (Placebo Comparator): Matching placebo to the phenazopyridine hydrochloride tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenazopyridine Hydrochloride — Tablets, 200 mg, every 8 hours for 48 hours.
  Other Names: Pyridium
  Arms: Phenazopyridine Hydrochloride Tablets, USP 200 mg
Drug: Placebo — Tablets, every 8 hours for 48 hours
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of Phenazopyridine Hydrochloride Tablets, USP 200 mg as a short term analgesic treatment for the primary symptoms of pain or burning when passing urine associated with uncomplicated urinary tract infections (uUTI)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncomplicated urinary tract infection (uUTI)
* Must have one of the following uUTI diagnosis
* Cystitis
* Urethritis
* A Positive urine dipstick test showing nitrate or leukocyte esterase (LE)
* Negative pregnancy test (if applicable)
* Must have one or both of the following symptoms of
* pain upon urination
* burning upon urination
* In addition, one of the following symptoms
* Not being able to empty bladder completely
* Pain or discomfort in lower abdomen, or pelvic areas
* Frequent urge to urinate
* Blood in urine
* None

Exclusion Criteria:

* Any diagnosis of a urinary tract or kidney disorder that is not a uUTI
* A diagnosis of Pyelonephritis (kidney infections when lower uUTI spreads to the upper tract)
* Women with a history of prior use of phenazopyridine hydrochloride
* Women who have taken any systemic anti-infectives within seven days of study participation
* Women with a history of G-6-PD deficiency or hemolytic anemia
* Women who have a known history of anatomical genitourinary (GU) anomalies or GU surgery within the past 6 months
* Women of child bearing age who do not consent to a pregnancy test
* Women who are lactating
* Chronic infection of the urinary tract requiring an intravenous pyelogram (IVP), ultrasound or cystoscopy
* Subjects with clinically significant abnormal results or finding on the screening physical examination, laboratory tests, vital signs or ECG.
* Subjects unable to comprehend the language of the informed consent and the self evaluation scales.
* Subjects with serious acute illness (e.g. pneumonia) or an untreated or unstable medical illness that would likely interfere with assessments of uUTI
* Subjects who have received an investigational medication as part of a drug trial 3 months prior to the baseline study visit
* Subjects with a history of severe drug allergy or hypersensitivity
* Subjects with a known sensitivity to Phenazopyridine, Hyoscyamine, Butabarbital and antibiotics.
* Employees of the investigator or the institution who have direct involvement in the trial or other trials under the direction of the investigator or their associates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
proportion of subjects in each treatment group who demonstrate reduction in pain or burning when passing urine. | 24 hrs after first dose and 48 hrs after second dose

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Pharmaceutical Resources, Inc., Totowa, New Jersey, United States